CLINICAL TRIAL: NCT03839810
Title: Effects of Stochastic Resonance Electrical Stimulation on Post Stroke Cortical Plasticity and Motor Function Recovery
Brief Title: Stochastic Resonance Stimulation in Brain Plasticity and Post Stroke Motor Recovery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Yang Ming Chiao Tung University (Other)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MOST107-2314-B-010-050
Record Dates: First submitted 2019-01-17; First posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Stroke, Ischemic; Healthy
Keywords: stochastic resonance; proprioception; motor control; motor recovery
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stochastic resonance (Experimental): stochastic resonance electrical stimulation is applied to the upper extremity during the subjects perform upper extremity motor function.
  Interventions: Other: stochastic resonance electrical stimulation
- sham stimulation (Sham Comparator): sham electrical stimulation (same electrode location, but no electrical current is applied) is applied to the upper extremity during the subjects perform upper extremity motor function.
  Interventions: Other: stochastic resonance electrical stimulation

INTERVENTIONS:
Other: stochastic resonance electrical stimulation — stochastic resonance electrical stimulation is applied in the upper extremity during motor functional training.
  Sham comparator group uses sham stimulation - same electrode location, but no electrical current is applied during motor functional training

SUMMARY:
This study evaluates the effectiveness of stochastic resonance electric stimulation on neuromuscular control and proprioception in healthy and individuals with stroke.

DETAILED DESCRIPTION:
Stroke is one of the leading causes of motor disability. The main intervention strategy in stroke rehabilitation is to induce cortical plasticity for motor re-learning.

It has been demonstrated that electrical stimulation applied to the periphery can elicit abundant sensory afferent inputs to enhance excitability and activation area in the sensorimotor cortex. Recent evidence suggested that a new type of electrical stimulation pattern, stochastic resonance stimulation, is capable of efficiently enhancing the activation of peripheral and central nervous system. Therefore, the purpose of this study are to identify the effects of stochastic resonance electrical stimulation on neuromuscular control and proprioception, and to investigate the effectiveness of combining stochastic resonance electrical stimulation with rehabilitation program on post stroke motor function recovery.

ELIGIBILITY:
In first stage

Inclusion Criteria:

healthy adults without history of neurological disorders or limitation in range of motion for thumb ﬂexion

In the second stage

Inclusion Criteria:

1. first-ever cerebral cortical region involved chronic stroke, onset over a month
2. able to perform active grasp on the affected side with the scores of manual muscle test at least two points
3. at stable medical condition for intervention confirmed by a specialized physician.

The exclusion criteria were

1. history of other neurological disorders
2. cognitive impairment (Mini-Mental State Examination score < 24, MMSE)29
3. unable to follow instructions
4. contraindications of ES
5. under 20 years old.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
EEG | baseline and one minute after stimulation
  we will calculate power spectral and see whether change in the alpha, beta, theta band
Fugl-Meyer Assessment for Upper Extremity | baseline and one minute after stimulation
  changes in upper extremity function of the stroke subjects

SECONDARY OUTCOMES:
force deviation | baseline and one minute after stimulation
  we first calculated the absolute value of the difference between force output and the value of 50%MVC for each data point and then calculated the average force deviation value by dividing the sum of all values by the number of data points
joint angle | baseline and one minute after stimulation
  ABS(the subject perform degree - target degree )
muscle activation | baseline and one minute after stimulation
  EMG changes in stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Li-Wei Chou, PhD, Principal Investigator — National Yang Ming Chiao Tung University
Locations (1):
- National Yang-Ming University, Taipei, Taiwan